CLINICAL TRIAL: NCT04219982
Title: A Randomized, Double-Blind Placebo-Controlled Phase 3 Study of the Safety, Pharmacokinetics, and Efficacy of DPI 386 Nasal Gel for the Prevention of Nausea Associated With Motion Sickness
Brief Title: DPI 386 Nasal Gel for the Prevention of Nausea Associated With Motion Sickness
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Failure to meet enrollment
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: DPI-386-07
Record Dates: First submitted 2019-03-11; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Intervention Model Description: The sample size of 54 allows for an equal distribution of subjects within gender and treatment arm: 18 subjects per treatment arm with 9 per gender.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is double-blinded for the DPI-386 Nasal Gel and placebo nasal gel arms. All DPI-386 Nasal Gel and placebo nasal gel vials are opaque and indistinguishable. The DPI-386 Nasal Gel and placebo nasal gel are identical in color and viscosity, and without identifiable smell.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DPI-386 Nasal Gel (Experimental): Active DPI-386 Nasal Gel
  Interventions: Drug: DPI-386 Nasal Gel
- DPI-386 Placebo Nasal Gel (Placebo Comparator): Placebo Nasal Gel
  Interventions: Drug: DPI-386 Placebo Nasal Gel
- Transderm Scop® (TDS) (Active Comparator): FDA approved Transderm Scop® (TDS).
  Interventions: Drug: Transderm Scop®

INTERVENTIONS:
Drug: DPI-386 Nasal Gel — Nasal gel
  Arms: DPI-386 Nasal Gel
Drug: DPI-386 Placebo Nasal Gel — DPI-386 Placebo Nasal Gel
  Arms: DPI-386 Placebo Nasal Gel
Drug: Transderm Scop® — Transderm Scop®
  Arms: Transderm Scop® (TDS)

SUMMARY:
Determine the efficacy, in terms of time to nausea (inclination to vomit), of DPI-386 Nasal Gel as compared to the current standard of care (TDS) and placebo nasal gel. • Describe the pharmacokinetics (PK) of a multi-dose schedule of DPI-386 Nasal Gel (0.2 mg twice a day for six consecutive days) as compared to the current standard of care (TDS). Determine the safety of a multi-dose schedule of DPI-386 Nasal Gel with an emphasis on cognitive adverse events as compared to the current standard of care (TDS) and placebo nasal gel. Determine how alertness is affected by administration of DPI-386 Nasal Gel, as compared to the current standard of care (TDS) and placebo nasal gel.

DETAILED DESCRIPTION:
Each subject eligible for the study on Day 0 will be assigned a subject number (starting with 101 for male subjects and 201 for female subjects) in consecutive order which will randomize the subject to one of the three study arms: double-blind DPI-386 Nasal Gel; double-blind placebo nasal gel; or Transderm Scop® (TDS). The subject number will link the nasal gel (active or placebo) treatment arms (double-blind) to a multi digit random number (study drug kit number) different from the subject number. The nasal gel vials, contained in the study drug kit, will be labelled with the same study drug kit number. Each 0.12 gram of the gel contains 0.2 mg of scopolamine HBr as the active ingredient along with the excipients sodium citrate, citric acid, sodium metabisulfite, glycerin, benzalkonium chloride, polyvinyl alcohol, and purified water.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated ICD.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 to 59 (inclusive).
4. Active duty military, reserves on active status, or dependents covered by Tricare health insurance. All potential subjects must be able to provide a current military or DoD dependent ID to be viewed by the PI or qualified designee prior to signing the ICD.
5. At least minimally susceptible to provocative motion as evidenced by a minimum score of 3.0 on the Motion Sickness Susceptibility Questionnaire (MSSQ).
6. In good general health as evidenced by medical history with no recent history or current diagnosis of clinical problems that would affect rotation in a vestibular study (e.g., vestibular pathology, seizure disorder, sinus congestion), as assessed by the PI or qualified designee.
7. Laboratory test results that are determined by the PI or qualified designee to be normal or - if slightly out of the normal range - determined to be not clinically significant. The following laboratory tests will be performed:

   1. Hematology panel (WBC, RBC, HGB, Hct)
   2. Biochemistry panel (liver function: bilirubin [total and direct], ALT, AST, ALP, and GGT; Albumin, Creatinine, BUN, and Cortisol)
   3. Electrolytes (Na+, K+, Cl-, Ca2+, and PO4)
8. Ability to take intranasal medication and willingness to adhere to the study schedule and time constraints.
9. For females of child-bearing potential: willingness to provide a urine sample for the hCG pregnancy test upon every visit to NAMRU-D. Test must be negative.
10. Agreement to adhere to the following lifestyle considerations:

    1. Refrain from consumption of grapefruit and any substance containing grapefruit for seven days prior to, during, and for seven days after the six treatment days.
    2. Caffeine intake limited to 900 mg per day (six 8-ounce cups per day [daily total of 1.4 liters]) during the six treatment days.
    3. Abstain from alcohol for 24 hours prior to first dose of study medication and during the six treatment days.
    4. Cigarettes limited to no more than one pack per day; cigars to one per day; and chewing tobacco to no more than a quarter of a can per day during the six treatment days.

Exclusion Criteria:

* 1. Pregnancy, lactation, or positive urine pregnancy test at screening.

  2. Known allergic reactions to scopolamine or other anticholinergics.

  3. Currently prescribed any of the following medication types: belladonna alkaloids, antihistamines (including meclizine), tricyclic antidepressants, muscle relaxants and nasal decongestants.

  4. Hospitalization or significant surgery requiring hospital admittance within the past six months.

  5. Treatment with another investigational drug or other intervention within the past 30 days.

  6. Having donated blood or plasma or suffered significant blood loss within the past 30 days.

  7. Use of a nicotine patch. 8. Having any of the following medical conditions within the last two years or if any of the following medical conditions were experienced more than two years ago and are deemed clinically significant by the PI or qualified designee:
  1. Significant gastrointestinal disorder, asthma, or seizure disorders.
  2. History of vestibular disorders.
  3. History of narrow-angle glaucoma.
  4. History of urinary retention.
  5. History of alcohol or drug abuse.
  6. Nasal, nasal sinus, or nasal mucosa surgery.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
The length of time spent in mechanical rotation until nausea (inclination to vomit) is achieved, or 20 minutes have elapsed. | up to 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David Helton, Study Director — Repurposed Therapeutics, Inc.
Locations (1):
- NAMRU-D, Dayton, Ohio, United States